CLINICAL TRIAL: NCT06763133
Title: The Effect of Cold Water Spray Application on Dry Mouth and Thirst Symptoms and Comfort of Patients After Endonasal Endoscopic Surgery After Admission to Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Didem Özdağ, Registered Nurse, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SaglikBilimleriU-SBF-DO-01
Record Dates: First submitted 2024-12-23; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Thirst in Intensive Care Unit (ICU) Practice; Thirst; Due to Deprivation of Water; Thirst; Dry Mouth; Comfort
Keywords: Endonasal Endoscopic Surgery; Postoperative Nursing; Thirst; Cold Water; Spray; Oral Care; Comfort; Nose Tampon
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: Patient groups Experimental Group: Patients in this group will receive cold water application in the form of a spray (6 times every half hour) and oral care (2 times a day, at 22.00 pm and 07.00 am, using an oral care solution containing 0.25% chlorhexidine gluconate approved by the Ministry of Health and an oral care stick, and moisturizing the lips with a lip moisturizer containing glycerin as the main component).
  Control Group: Patients in this group will be given 2 cc of water at room temperature into the patient's mouth with the syringe routinely applied for mouth wetting in the clinic (1 time every hour) and oral care (2 times a day, at 22:00 in the evening and 07:00 in the morning, using oral care solution containing 0.25% chlorhexidine gluconate approved by the Ministry of Health and oral care stick, and moisturizing the lips with lip moisturizer with glycerin as the main component).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Patients in this group will receive cold water application in the form of a spray (6 times every half hour) and oral care (2 times a day, at 22.00 pm and 07.00 am, using an oral care solution containing 0.25% chlorhexidine gluconate approved by the Ministry of Health and an oral care stick, and moisturizing the lips with a lip moisturizer containing glycerin as the main component).
  Interventions: Other: Cold Water Spray Application
- Control Group (Other): Patients in this group will be given 2 cc of water at room temperature into the patient's mouth with the syringe routinely applied for mouth wetting in the clinic (1 time every hour) and oral care (2 times a day, at 22:00 in the evening and 07:00 in the morning, using oral care solution containing 0.25% chlorhexidine gluconate approved by the Ministry of Health and oral care stick, and moisturizing the lips with lip moisturizer with glycerin as the main component).
  Interventions: Other: Clinical routine practice

INTERVENTIONS:
Other: Cold Water Spray Application — Cold water spray application after endonasal endoscopic surgery.
  Arms: Experimental Group
Other: Clinical routine practice — The process of giving 2 cc of water to patients with a syringe as a clinical routine practice.
  Arms: Control Group

SUMMARY:
The aim of this observational study was to evaluate the effect of cold water spray application on dry mouth and thirst symptoms and comfort of patients who underwent endonasal endoscopic pituitary surgery in neurosurgery in the first 24 hours after admission to intensive care unit.

The main questions it aims to answer are as follows:

H0.1: Cold water spray application has no effect on dry mouth symptoms. H1.1: The cold water spray application has an effect on the dry mouth symptom. H0.2: The cold water spray application has no effect on the thirst symptom. H1.2: Cold water spray application has an effect on thirst symptom. H0.3: Cold water spray application has no effect on oral health. H1.3: Cold water spray application has an effect on oral health. H0.4: Cold water spray application has no effect on patient comfort. H1.4: Cold water spray application has an effect on patient comfort. The research sample will be divided into two as treatment and control groups. A web-based random sample selection will be made to determine the patients to be included in the research groups. Cold water spray will be applied to the treatment group and their data will be recorded. Clinical routine will continue to be applied to the control group.

DETAILED DESCRIPTION:
The endoscope has been used in surgery for many years due to the favorable factors such as small incision area. In the 1990s, the experience gained in surgery and advances in technology were adapted to endoscopy and new endoscopic approaches were developed in transsphenoidal surgery. Although this method varies according to the type of surgical procedure, the nature and localization of the mass and the decision of the surgeon, it is a method that is now used in neurosurgery.

Studies have shown that pain, various pulmonary, cardiovascular and neurologic symptoms, deterioration in stability, anxiety, nausea and vomiting, insomnia, limitation of movement, thirst and dry mouth are the most common issues that patients experience after surgery. In endonasal endoscopic surgery, preoperative fluid and nutrient restriction and anxiety, intraoperative anesthetic drugs, intubation, surgical procedure, postoperative neuroendocrine response to surgical stress, hormonal irregularities due to pituitary surgery, fluid-electrolyte imbalances, and the tampon placed to stabilize the graft placed between the nose and skull base after the surgical procedure can cause patients to experience severe dry mouth and thirst. These tampons used for graft stabilization can remain in the patient for an average of 5-7 days. This may cause patients to experience more thirst and dry mouth symptoms.

When the literature is examined, it is seen that thirst and dry mouth symptoms experienced by patients and the effectiveness of the interventions have been evaluated in recent years. However, there is no study evaluating thirst and dry mouth symptoms in patients undergoing endonasal endoscopic surgery. It is thought to be important to evaluate the effectiveness of cold water spray application on dry mouth and thirst symptoms, which are thought to affect the comfort levels of patients in this patient group.

Hypotheses of the Study H0.1: Cold water spray application has no effect on dry mouth symptom. H1.1: Cold water spray application has an effect on dry mouth symptom. H0.2: The cold water spray application has no effect on the thirst symptom. H1.2: Cold water spray application has an effect on thirst symptom. H0.3: Cold water spray application has no effect on oral health. H1.3: Cold water spray application has an effect on oral health. H0.4: Cold water spray application has no effect on patient comfort. H1.4: Cold water spray application has an effect on patient comfort. Inclusion criteria

* Patients who agreed to participate in the study,
* Patients over 18 years of age,
* Patients with endonasal endoscopic surgery and nasal tampons,
* Patients who can communicate verbally,
* Patients with a Glasgow Coma Scale score of 15 before and after surgery. Exclusion criteria
* Patients who refused to participate in the study,
* Patients under 18 years of age,
* Patients who require respiratory support after surgical intervention and need intubation,
* Patients undergoing surgery that may interfere with oral assessment,
* Patients with a postoperative Glasgow Coma Scale score of 14 or less,
* Patients with Diabetes Mellitus and Xerostomia. Patient groups Experimental Group: Patients in this group will receive cold water application in the form of a spray (6 times every half hour) and oral care (2 times a day, at 22.00 pm and 07.00 am, using an oral care solution containing 0.25% chlorhexidine gluconate approved by the Ministry of Health and an oral care stick, and moisturizing the lips with a lip moisturizer containing glycerin as the main component).

Control Group: Patients in this group will be given 2 cc of water at room temperature into the patient's mouth with the syringe routinely applied for mouth wetting in the clinic (1 time every hour) and oral care (2 times a day, at 22:00 in the evening and 07:00 in the morning, using oral care solution containing 0.25% chlorhexidine gluconate approved by the Ministry of Health and oral care stick, and moisturizing the lips with lip moisturizer with glycerin as the main component).

Primary Objective of the Study (Postoperative 1.2.4.8 and 24th hour within the first 24 hours postoperatively) To assess thirst status: A numerical rating scale numbered 0-10, 0: no thirst, 10: unbearable thirst (1-3 mild, 4-6 moderate, 7-10 severe), will be used.

To assess dry mouth: Numeric rating scale numbered 0-10, 0: no dry mouth, 10: intolerable dry mouth (1-3 mild, 4-6 moderate, 7-10 severe), will be used.

To assess oral health: The Oral Health Assesment Tool will be used. The original scale consists of eight categories: lips, tongue, gums and mucosa, saliva, teeth, presence of dentures, oral cleanliness and toothache. The lowest score to be obtained from the scale is 0 and the highest score is 16. Scores can range from 0 - very healthy to 16 - very unhealthy. In this study, the first four items of the scale, 'lips, tongue, gums-mucosa and saliva' categories will be used. In this case, the lowest score to be obtained from the scale will be 0 and the highest score will be 8. The validity and reliability of the OHAT in Turkish has been established.

Secondary Objective of the Study (Postoperative 24th hour, when the patient leaves the intensive care unit) To determine the comfort level: Perianesthesia Comfort Scale will be used. The scale consists of 24 items developed to assess the patient's comfort before and after surgery. Each item in the scale has Likert-type scoring and has a score ranging from 1-6 from "Strongly Disagree" to "Strongly Agree". The highest total score that can be obtained from the scale is 144 and the lowest total score is 24. A low score indicates poor comfort, while a high score indicates good comfort. The Turkish validity and reliability study of the scale was conducted and Cronbach's alpha coefficient was found to be 0.83.

Research Flow Steps:

A. Preoperative;

1. After the surgical operation is decided and the patient is hospitalized in the clinic, the patient will be interviewed and informed about the study.
2. Consent will be obtained from patients who agree to participate in the study and a voluntary consent form will be signed.
3. Patient data will be collected using the 'Data Collection Form'.
4. The inclusion criteria of the patient who agrees to participate in the study will be evaluated.
5. The group in which the patient who meets the inclusion criteria will be included will be determined by web-based sample selection method.

B. Postoperative;

1. The level of consciousness, airway protection, nausea and vomiting status of the patient admitted to the intensive care unit after surgery will be evaluated with the help of the 'Safe Protocol for the Management of Early Postoperative Thirst' in order to prevent the risk of aspiration within the scope of patient safety.

3. Patients who meet the criteria will be started to be administered from the 1st hour after intensive care admission.

4. Patients who do not meet the criteria will be evaluated regularly every half hour and the intervention will be started after airway safety is ensured.

5. Patients in the application group;

a) The vital signs, pain score, presence of nausea and vomiting, Glasgow score, thirst and dry mouth scores, OHAT scores of the patients will be evaluated and recorded at 1.2.4.8 and 24 hours.

b) Cold water spray, which is kept in 30 cc plastic bottles at +4 degrees in the refrigerator, will be sprayed into the patient's mouth 6 times every half hour, corresponding to 1 cc.

c) Oral status of the patients will be evaluated using the OHAT scale at 1.2.4.8 and 24 hours postoperatively.

d) Patient oral care will be performed twice a day, at 22.00 pm and 07.00 am, using oral care solution containing 0.25% chlorhexidine gluconate approved by the Ministry of Health, using an oral care stick, and moisturizing the lips with lip moisturizer with glycerin as the main component.

6. Patients in the control group;

1. Vital signs, pain score, presence of nausea and vomiting, Glasgow score, thirst and dry mouth scores, OHAT scores will be evaluated and recorded at 1.2.4.8 and 24 hours.
2. 2 cc water at room temperature, which is a clinical routine practice, will be given to the patient every hour with the help of a syringe.
3. Oral status of the patients will be evaluated using the OHAT scale at 1.2.4.8 and 24 hours postoperatively.
4. Patient oral care will be performed twice a day, at 22.00 pm and 07.00 am, using oral care solution containing 0.25% chlorhexidine gluconate approved by the Ministry of Health, using an oral care stick, and moisturizing the lips with lip moisturizer with glycerin as the main component.

   7. In order to protect the circadian rhythms of the patients, applications will not be performed between 00:00-06:00.

   8. Patient comfort will be evaluated using the 'Perianesthesia Comfort Scale' when the patient leaves the intensive care unit at the 24th postoperative hour.

   9. Data will be collected from patients at 1, 2, 4, 8 and 24 hours postoperatively.

   The study is planned to be conducted between January 2024 and December 2024 among patients who underwent endonasal endoscopic surgery in the Neurosurgery Clinic of Ankara Gülhane Training and Research Hospital. Power analysis was performed using G-power 3.1.3 software package to calculate the required number of patients. Based on a study conducted by Öztaş and Öztaş, it was determined that 32 patients were needed to determine the effect size of 1.20 with 90% power. Statistically, the significance level was determined as 0.05. Since it was thought that there might be data loss, the number of patients in the groups was determined as 20 with 10% more people. A web-based random sample selection will be conducted to determine the patients to be included in the research groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agreed to participate in the study,
* Patients over 18 years of age,
* Patients with endonasal endoscopic surgery and nasal tampons,
* Patients who can communicate verbally,
* Patients with a Glasgow Coma Scale score of 15 before and after surgery.

Exclusion Criteria:

* Patients who refused to participate in the study,
* Patients under 18 years of age,
* Patients who require respiratory support after surgical intervention and need intubation,
* Patients undergoing surgery that may interfere with oral assessment,
* Patients with a postoperative Glasgow Coma Scale score of 14 or less,
* Patients with Diabetes Mellitus and Xerostomia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Feeling of Thirst and Dry Mouth Experienced by Patients in the First 24 Hours After Surgery | Within the first 24 hours postoperatively, evaluations will be made at the 1st, 2nd, 4th, 8th and 24th hours.
  To assess thirst status, a numerical assessment scale numbered 0-10 will be used, where 0: no thirst, 10: unbearable thirst (1-3 mild, 4-6 moderate, 7-10 severe).
  To assess dry mouth: a numerical rating scale numbered 0-10 will be used, where 0: no dry mouth, 10: unbearable dry mouth (1-3 mild, 4-6 moderate, 7-10 severe).
  The Oral Health Assesment Tool will be used to assess oral status. The original scale consists of eight categories: lips, tongue, gums and mucosa, saliva, teeth, presence of dentures, oral hygiene, and toothache. The lowest score to be obtained from the scale is 0, while the highest score is 16. Scores can vary between 0-very healthy and 16-very unhealthy. In this study, the first four items of the scale, which are 'lips, tongue, gums-mucosa, and saliva' categories, will be used. In this case, the lowest score to be obtained from the scale will be 0, while the highest score will be evaluated as 8. The validity and reliability of the OHAT in Turkish has been conducted

SECONDARY OUTCOMES:
Evaluation of Patient Comfort When Leaving the Intensive Care Unit After 24 Hours Postoperatively | At the end of the 24th postoperative hour, before the patient leaves the intensive care unit
  To determine the comfort level: Perianesthesia Comfort Scale will be used. The scale consists of 24 items developed to evaluate the patient's comfort before and after surgery. Each item in the scale has a Likert-type scoring system and has a score ranging from 1-6 from "Strongly Disagree" to "Strongly Agree". The highest total score that can be obtained from the scale is 144, and the lowest total score is 24. A low score indicates poor comfort, a high score indicates good comfort. The scale's Turkish validity and reliability study was conducted and Cronbach's alpha coefficient was found to be 0.83.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I want to decide after I finish my thesis.